CLINICAL TRIAL: NCT02154594
Title: "The Efficacy of Acacia Catechu Mouthrinse as Antiplaque and Antigingivitis Agent in Fixed Orthodontic Appliance Patients.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tatyasaheb Kore Dental College (Other)
Responsible Party: Principal Investigator, DR.DHANASHREE RAVINDRA AGARWAL, POST GRADUATE STUDENT IN PERIODONTOLOGY, Tatyasaheb Kore Dental College
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: DHANASHREE289
Record Dates: First submitted 2014-05-26; First posted 2014-06-03 (Estimated); Last update posted 2014-06-03 (Estimated); Status verified 2014-05

CONDITIONS: Gingivitis
Keywords: Acacia; Chlorhexidine; Gingivitis; Orthodontic appliances.
MeSH Terms: conditions — Gingivitis | interventions — chlorhexidine gluconate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Acacia (Experimental): Rinse with 20 ml of Acacia catechu mouthwash twice daily for 15 days
  Interventions: Drug: Acacia catechu; Drug: Chlorhexidine gluconate; Other: Distilled water
- Chlorhexidine gluconate (Active Comparator): Rinse with 10 ml of chlorhexidine mouthwash twice daily for 15 days
  Interventions: Drug: Acacia catechu; Drug: Chlorhexidine gluconate; Other: Distilled water
- Distilled water (Placebo Comparator): Rinse with 10 ml distilled water twice daily for 15 days.
  Interventions: Drug: Acacia catechu; Drug: Chlorhexidine gluconate; Other: Distilled water

INTERVENTIONS:
Drug: Acacia catechu
Drug: Chlorhexidine gluconate
  Other Names: Hexidine
Other: Distilled water

SUMMARY:
To study effect of acacia catechu a herbal extract;as antipaque and antigingivitis agent in patients with fixed orthodontic appliances.This study is a double blind randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* 60 patients in the age group of 15-30 yrs
* plaque induced gingivitis having fixed orthodontic appliance

Exclusion Criteria:

* seeking any type of antibacterial mouthwash within four weeks of commencement of study,
* history of any systemic disease, or past illness,
* mentally or physically handicapped,
* history of smoking, tobacco chewing, alcohol consumption,
* patients with periodontitis, pregnant and lactating women

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2014-02; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in Plaque index(PI) | 15 Days

SECONDARY OUTCOMES:
Changes from baseline in Gingival index(GI) | 15 Days

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Dhanashree R. Agarwal, B.D.S., Principal Investigator — Tatyasaheb Kore Dental College and Research Centre
Locations (1):
- Tatyasaheb Kore Dental College and Research Centre, Kolhāpur, Maharashtra, India